CLINICAL TRIAL: NCT00587717
Title: The Acute Effect of Inflammatory Markers of Atherosclerotic Plaque in Humans
Brief Title: The Acute Effect of Statins on Inflammatory Markers of Athersclerotic Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Amir Lerman, M.D. (principal investigator, Mayo clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 485-02; Merck #02005
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Carotid Artery Disease
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Two 80 mg pills simvastatin taken 24 hours prior to surgery
  Interventions: Drug: simvastatin
- 2 (Placebo Comparator): Two 80 mg pills placebo are taken 24 hours prior to surgery
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: simvastatin — Two 80 mg pills simvastatin taken 24 hours prior to surgery
  Other Names: Zocor
  Arms: 1
Drug: placebo — take 2 80 mg pills placebo 24 hours prior to surgery
  Arms: 2

SUMMARY:
This study is being done to determine if the acute administration of the drug Simvastatin reduces plaque tissue inflammation and plaque instability in patients undergoing carotid endarectomy

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing carotid endarterectomy
* No previously known side effects of statins
* Patients who will sign an informed consent
* Age > 18 years old
* No signs of current infection

Exclusion Criteria:

* Patient hypersensitive to any component of this medication
* Patients with acute liver disease (AST> normal value)
* Patients with chronic liver disease (history of Hepatitis B or C)
* Patients with renal failure (creatinine > 3.0)
* Patients with unexplained muscle pains and aches
* Patients with rheumatoid arthritis
* Patients with Lupus
* Current cancer treatment
* Patients on cyclosporin, digoxin, Itraconazole, Ketoconazole and other antifungal azoles, the macrolide antibiotics and antidepressant nefazodone
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2002-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
This study is being done to see if giving the study drug, Simvastatin, quickly lessens the swelling of plaque tissue (tissue around your heart) and plaque movement in patients undergoing cqrotid endarterectomy procedure. | 24 prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic